CLINICAL TRIAL: NCT02071745
Title: Navigated Total Knee Arthroplasty, the Correlation to CT Scans and Clinical Results
Status: Completed | Type: Observational
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, David Eliya Rothem, MD, Ziv Hospital
Other Study IDs: ZIV-0041-13
Record Dates: First submitted 2014-02-18; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Navigation

SUMMARY:
Total knee replacement is one of the most commonly performed orthopedic procedures. As of 2010, about 600,000 total knee replacements were being performed annually in the United States and these numbers are rising. The normal knee joint functions as a complex hinge allowing primarily ﬂexion and extension, rotation and gliding. The knee joint is made up of three compartments, the lateral, medial and anterior (patellofemoral). Damage to the cartilage of one or more compartments may be the result of osteoarthritis (idiopathic or post-traumatic), inﬂammatory arthritis (rheumatoid,psoriatic, etc.), a-vascular necrosis, tumors, or congenital deformities. Osteoarthritis and rheumatoid arthritis are the causes of the overwhelming majority of total joint arthroplasties.

A successful Total knee arthroplasty(TKA) surgery includes: an accurate alignment( the mechanical axis in axial and rotational planes), as well as significant pain relief which improves function and quality of life. Incorrect alignment can lead to abnormal wear, premature mechanical loosening of the components and patellofemoral problems.

The common techniques for Total knee replacement are:

1. Conventional method TKR
2. CT/MRI-based preoperative navigated TKR
3. Image-free intraoperative navigated TKR In our research we focus on the 3rd method using the Orthopilot navigation system Aesculap®, Tutlingen, Germany. This system is an active PC based guiding system that helps the surgeon decide on the accurate alignment and orientation of the implant and cutting surfaces of the bone and thus avoid incorrect alignment.

We aim to compare between pre-operative and post-operative lower limb alignment (mechanical axis) in Aesculap based TKA using serview CT. Furthermore, we will try to examine the existence of a correlation between the CT scans and the Orthopilot navigation system output and assess the clinical outcome of the patient postoperatively.

Our Hypothesis is that the intra-operative navigation system is accurate and correlated to CT images results, moreover, allows the surgeon to achieve a good mechanical axis and high clinical outcome,

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* severe osteoarthrosis of the knee
* failure of conservative treatment.

Exclusion Criteria:

* patients with severe vascular disease
* secondary knee deformation due to muscular atrophy or disease
* active infection
* morbid obesity
* neuropathic knee and osteomyelitis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing navigated total knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
limb axis measurement | An average, 1 week preoperatively up to 3 days postoperatively.
  surview CT images pre-( 1 week before the operation) and post-operatively(the day of operation) will be analyzed using the Traumacad software for limb axis.
  The navigation system results pre- and post-operatively will be given by the computer as an output at the Operation Theater.
  The results will be recorded for Varus/Valgus and degrees of deformity.

SECONDARY OUTCOMES:
Clinical outcome and function | up to 6 months postoperatively
  the clinical evaluation of the patient will be based on the knee society scoring system: Range of movement(degrees), pain level(1-lowest,10-highest), anterior-posterior stability(mm), mediolateral stability(degrees), function test based on walking,climbing stairs, use of walking aids. The results will be summed up and give a numerical score.

CONTACTS AND LOCATIONS:
Overall Officials: David E Rothem, MD, Principal Investigator — Head of joint repalcement unit, Orthopedic department, Ziv medical center, Safed, Israel
Locations (1):
- ZIV medical center, Safed, Israel

REFERENCES:
- [Result] Mason JB, Fehring T, Fahrbach K. Navigated total knee replacement. J Bone Joint Surg Am. 2007 Nov;89(11):2547-8; author reply 2548; discussion 2548-50. doi: 10.2106/00004623-200711000-00032. No abstract available. PMID 17974899
- [Result] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Result] Oswald MH, Jakob RP, Schneider E, Hoogewoud HM. Radiological analysis of normal axial alignment of femur and tibia in view of total knee arthroplasty. J Arthroplasty. 1993 Aug;8(4):419-26. doi: 10.1016/s0883-5403(06)80042-2. PMID 8409995
- [Result] Wasielewski RC, Galante JO, Leighty RM, Natarajan RN, Rosenberg AG. Wear patterns on retrieved polyethylene tibial inserts and their relationship to technical considerations during total knee arthroplasty. Clin Orthop Relat Res. 1994 Feb;(299):31-43. PMID 8119035
- [Result] Bargren JH, Blaha JD, Freeman MA. Alignment in total knee arthroplasty. Correlated biomechanical and clinical observations. Clin Orthop Relat Res. 1983 Mar;(173):178-83. PMID 6825330
- [Result] Berger RA, Rubash HE, Seel MJ, Thompson WH, Crossett LS. Determining the rotational alignment of the femoral component in total knee arthroplasty using the epicondylar axis. Clin Orthop Relat Res. 1993 Jan;(286):40-7. PMID 8425366
- See also: Related Info — http://www.ahrq.gov/data/hcup/